CLINICAL TRIAL: NCT01080664
Title: A Phase I, Dose-escalation Study of AS703569 Given Orally to Subjects With Haematological Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Please see Purpose Statement below
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27335
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Haematological Malignancies
Keywords: AS703569; Aurora Kinase Inhibitor; Haematological malignancies
MeSH Terms: interventions — MSC1992371A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen 1 (Experimental): Regimen 1: AS703569 administered on Days 1, 2, 3 and Days 8, 9, 10 of a 21-day cycle
  Interventions: Drug: AS703569
- Regimen 2 (Experimental): Regimen 2: AS703569 administered on Days 1, 2, 3, 4, 5, 6 of a 21-day cycle
  Interventions: Drug: AS703569

INTERVENTIONS:
Drug: AS703569 — Dose Escalation
  Regimen 1 - 3-47 mg/m2/day, orally once daily on days 1, 2,3 and 8, 9, 10 of a 21 day cycle:
  Number of cycles: until progression or unacceptable toxicity develops.
  Cohort Expansion
  Regimen 1 - Maximum tolerated dose from dose-escalation part or a lower dose in mg/m2/day, orally once daily on days 1, 2,3 and 8, 9, 10 of a 21 day cycle:
  Number of cycles: until progression or unacceptable toxicity develops
  Other Names: Aurora kinase inhibitor
  Arms: Regimen 1
Drug: AS703569 — Dose Escalation Regimen 2 - 3-47 mg/m2/day, orally once daily on days 1, 2, 3, 4, 5, 6 of a 21 day cycle Number of cycles: until progression or unacceptable toxicity develops.
  Cohort Expansion Regimen 2 - Maximum tolerated dose from dose-escalation part or a lower dose in mg/m2/day, orally once daily on days 1, 2, 3, 4, 5, 6 of a 21 day cycle Number of cycles: until progression or unacceptable toxicity develops.
  Other Names: Aurora kinase inhibitor
  Arms: Regimen 2

SUMMARY:
EMD Serono decided to terminate enrollment based on a review of the available clinical data and low probability of completing the trial based on the observed recruitment rate. Subjects already enrolled in the study continued participation in the study, consistent with the protocol, to study completion.

DETAILED DESCRIPTION:
The goal of this research study is to investigate for the first time the safety and tolerability of a new drug (AS703569), called an aurora kinase inhibitor, being tested to treat blood cancers in patients with different blood cancers. The research study will also assess how the body breaks down AS703569 and what changes occur in the blood after oral doses of AS703569. It will also look to see if there is any improvement in your blood cancer. The use of AS703569 in this study is experimental.

ELIGIBILITY:
Inclusion Criteria:

Dose-escalation part:

* Primary or secondary acute myeloid leukaemia, including subjects:

with first or subsequent relapse after standard therapy, with no established treatment options; refractory to available therapies, e.g. who failed to achieve complete remission after chemotherapies; Newly-diagnosed elderly subjects (over 60 years) according to WHO classification (≥20 blasts in bone marrow), who did not accept or were not eligible for chemotherapy (first line therapy)

* Subjects with myelodysplastic syndrome (IPSS Int-2 or high risk) resistant or intolerant to standard treatment and not candidates for allogeneic HSCT.
* Subjects with chronic myeloid leukaemia in chronic, accelerated or blast-phase, resistant or intolerant to standard treatment and not candidates for allogeneic HSCT.
* Subjects with myeloproliferative disorders and no effective treatment options.
* Subjects with acute lymphoblastic leukaemia, relapsing, resistant or intolerant to standard treatment and no effective treatment options.
* Subjects with chronic lymphocytic leukaemia, relapsing, resistant or intolerant to standard treatment and no effective treatment options.
* Subjects with non-Hodgkin lymphoma, relapsing, resistant or intolerant to standard treatment with no effective treatment options.

Cohort expansion part

* Primary or secondary acute myeloid leukaemia not eligible for chemotherapy (first line therapy), including subjects

with first or subsequent relapse after standard therapy, for whom no established treatment options are available; refractory to available therapies, e.g. who failed to achieve complete remission after chemotherapies; Newly-diagnosed elderly subjects (over 60 years) according to WHO classification (≥ 20 blasts in bone marrow), who did not accept or were not eligible for chemotherapy (first line therapy)

* Subjects with chronic myeloid leukaemia in chronic or accelerated phase, resistant or intolerant to standard treatment, who have not achieved a complete haematological response, and are not candidates for allogeneic HSCT.
* Subjects with myeloproliferative disorders with no effective treatment options.
* Subjects with Philadelphia chromosome positive acute leukaemias including acute lymphoblastic leukaemia and blast phase chronic myeloid leukaemia, relapsing, resistant or intolerant to standard treatment with no effective treatment options.

Exclusion Criteria:

* Acute promyelocytic leukaemia.
* Ongoing uncontrolled bacterial, viral, fungal or atypical mycobacterial infection.
* Hyperleukocytosis with >50x10(9)/L leukaemic blasts.
* Chemotherapy, immunotherapy, biologic therapy or any experimental anti-cancer therapy within 28days prior to study Day1 and/or not having recovered from its toxicity.
* Extensive radiotherapy involving ≥30% of bone marrow (e.g. whole pelvis, half spine) within 6months prior to study Day1.
* Active CNS disease involvement.
* Any condition, including laboratory, medical history or pre-study assessment findings, that in the opinion of the Investigator, constitute a risk or contraindication for participation or that could interfere with the study objectives, conduct or evaluation of a drug to be taken orally.
* Clinically relevant cardiac abnormalities or clinically relevant abnormalities .
* Known infection with human immunodeficiency virus, active hepatitis B, or hepatitis C.
* Signs and symptoms suggestive of transmissible spongiform encephalopathy.
* Major surgery within 2weeks prior to study Day1.
* Haemoglobin <8g/dL at screening (can be transfused).
* Refractory to platelet transfusion (defined as increase of <20.109/L platelets 1hour after transfusion).
* Coexistent second malignancy or history of prior malignancy within previous 3years (excluding basal or squamous cell carcinoma of the skin, and in situ carcinoma of the cervix that has been treated curatively).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2006-12; Primary Completion 2010-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | 21 days or 1 cycle
  Dose-escalation part - The number of subjects experiencing at least a Dose-Limiting Toxicity (DLT), judged to be related to the study medication, evaluated over the first cycle only for each dose level and regimen, independently.
Preliminary anti-tumour activity | 42 days or 2 cycles
  Cohort expansion part - Preliminary anti-tumour activity in four selected cohorts of haematological malignancies as assessed every two cycles

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAE) | minimum 21 days or 1 cycle
  Dose-escalation and Cohort expansion parts The proportion/number of subjects experiencing treatment-emergent adverse events (TEAE) after the first cycle and during multiple cycles, in each cohort for each of the 2 dose-regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Narmyn Rejeb, M.D., Study Director — Merck Serono S.A., Geneva
Locations (10):
- CTRC at the UT Health Science Center at San Antonio, San Antonio, Texas, United States
- Belgium (2):
  - Haematologie UZ Gasthuisberg, Leuven
  - Mont-Godinne University Hospital (UCL), Yvoir
- Germany (3):
  - Universitatsklinik Frankfurt, Frankfurt am Main
  - Technische Universitat Munchen, München
  - Medizinische Universitatsklinik, Ulm
- Policlinico Sant'Orsola Malpighi, Bologna, Italy
- Switzerland (3):
  - Kantonsspital Basel, Basel
  - Hospitaux Universitaires, Geneva
  - Kantonsspital St Gallen, Sankt Gallen

REFERENCES:
- [Derived] Graux C, Sonet A, Maertens J, Duyster J, Greiner J, Chalandon Y, Martinelli G, Hess D, Heim D, Giles FJ, Kelly KR, Gianella-Borradori A, Longerey B, Asatiani E, Rejeb N, Ottmann OG. A phase I dose-escalation study of MSC1992371A, an oral inhibitor of aurora and other kinases, in advanced hematologic malignancies. Leuk Res. 2013 Sep;37(9):1100-6. doi: 10.1016/j.leukres.2013.04.025. Epub 2013 Jun 5. PMID 23746966